CLINICAL TRIAL: NCT04369014
Title: Characteristic Changes During Anesthesia With Etomidate and Propofol
Brief Title: Effect of Etomidate and Propofol on Electroencephalography
Acronym: CHAPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: XJH-A-20200330
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: General Anesthesia
Keywords: electroencephalography; etomidate; propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- etomidate (Experimental)
  Interventions: Drug: etomidate anesthesia
- propofol (Experimental)
  Interventions: Drug: propofol anesthesia

INTERVENTIONS:
Drug: etomidate anesthesia — etomidate is used for induction and maintenance of general anesthesia
  Arms: etomidate
Drug: propofol anesthesia — propofol is used for induction and maintenance of general anesthesia
  Arms: propofol

SUMMARY:
Electroencephalography (EEG) monitoring reflect the brain electro-activity. Different anesthetics may show different changes in EEG during anesthesia. Etomidate and propofol are widely used for general anesthesia. The characteristic changes of these two anesthetics may be different.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery under general anesthesia
* Patients provided written informed consent

Exclusion Criteria:

* Patients with history of neurological or psychiatric diseases
* Patients younger than 18 years old
* Patients scheduled for surgery involved head
* Patients with pregnancy or planned for breeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
delta wave deficiency during anesthesia | from anesthesia induction to extubation of the endotracheal tube, on an average of 2.5 hours

SECONDARY OUTCOMES:
spindle wave deficiency during anesthesia | from anesthesia induction to extubation of the endotracheal tube, on an average of 2.5 hours
burst suppression during anesthesia | from anesthesia induction to extubation of the endotracheal tube, on an average of 2.5 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No